CLINICAL TRIAL: NCT06318637
Title: A Clinical Evaluation of the Acceptability and Feasibility to Caregivers of a Bedtime Routine for Neonates
Brief Title: Evaluation of the Acceptability and Feasibility of a Bedtime Routine for Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCSSKB005432
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-06

CONDITIONS: Newborn
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will follow their typical daily activities with their baby throughout the study, including their typical bathing, skincare, and sleep practices.
  Interventions: Other: Daily Activities
- Interventional Group (Wash/Shampoo and Lotion) (Experimental): Participants in the intervention group will use the provided wash/shampoo, and face and body lotion for their baby. At Baseline, participants caregivers in the intervention group will be provided with instructions for institution of a daily bedtime routine for their infant, which includes a massage with a moisturizing lotion.
  Interventions: Other: Baby Wash/Shampoo; Other: Body Lotion

INTERVENTIONS:
Other: Baby Wash/Shampoo — Marketed baby wash/shampoo to be used as needed.
  Arms: Interventional Group (Wash/Shampoo and Lotion)
Other: Daily Activities — Participants to follow their typical daily activities with their baby.
  Arms: Control Group
Other: Body Lotion — Marketed body lotion to be used as needed.
  Arms: Interventional Group (Wash/Shampoo and Lotion)

SUMMARY:
The purpose of this study is to assess, via caregiver questionnaire, the acceptability and feasibility of implementing a bedtime routine for newborns.

ELIGIBILITY:
Inclusion Criteria:

Infant:

* Full term at birth (gestational age greater than or equal to [>=] 37 weeks)
* A singleton birth. (Having other infants/children in the household will be allowed but only 1 child per household may be enrolled)
* Breastfed, formula-fed, or combination

Caregiver:

* Able to read, write, speak, and understand English
* Must be the parent (biological or adoptive) and legal guardian of the infant participant who is willing and able to present proof of legal guardianship (example: birth certificate/hospital discharge paperwork along with valid ID of legal guardian, etc.)

Exclusion Criteria:

Caregiver and infant:

* Has known allergies or adverse reactions to common topical skincare products or the ingredients in the investigational study materials
* Has a history of or a concurrent health condition/situation which, in the opinion of the Principal Investigator (PI) or Study Physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other clinical study or has participated in a clinical study since infant's birth
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor
* Presents with a skin condition that may influence the outcome of the study (specifically psoriasis, eczema, atopic dermatitis, or erythema)

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Bedtime Routine Acceptability and Feasibility to Caregivers | At Day 10
  Will collect agreement data to statements on bedtime routine acceptability using a 5-point Likert scale, ranging from strongly agree to strongly disagree. Will collect bedtime routine information, including wash up/bath, massage/apply lotion and quiet activity.
Bedtime Routine Acceptability and Feasibility to Caregivers | At Day 17
  Will collect agreement data to statements on bedtime routine acceptability using a 5-point Likert scale, ranging from strongly agree to strongly disagree. Will collect bedtime routine information, including wash up/bath, massage/apply lotion and quiet activity.
Bedtime Routine Acceptability and Feasibility to Caregivers | At 3 months
  Will collect agreement data to statements on bedtime routine acceptability using a 5-point Likert scale, ranging from strongly agree to strongly disagree. Will collect bedtime routine information, including wash up/bath, massage/apply lotion and quiet activity.
Bedtime Routine Acceptability and Feasibility to Caregivers | At 6 months
  Will collect agreement data to statements on bedtime routine acceptability using a 5-point Likert scale, ranging from strongly agree to strongly disagree. Will collect bedtime routine information, including wash up/bath, massage/apply lotion and quiet activity.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rodgers, Ph.D., Principal Investigator — SGS North America, Inc.
Locations (1):
- SGS North America, Inc., Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu